CLINICAL TRIAL: NCT02509585
Title: A Prospective, Open-Label Trial of Comparing the Pathology Status of Lymphoseek®-Identified Sentinel Lymph Nodes Relative to the Pathological Pathology Status of Nonsentinel Lymph Nodes in Nodal Staging of Subjects With Known Cancer of the Cervix Who Are Undergoing Lymph Node Dissection
Brief Title: A Trial of Comparing the Pathology Status of Lymphoseek®-Identified Sentinel Lymph Nodes Relative to the Pathological Pathology Status of Nonsentinel Lymph Nodes in Nodal Staging of Subjects With Known Cancer of the Cervix Who Are Undergoing Lymph Node Dissection
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low accrual
Sponsor: Cardinal Health 414, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NAV3-19
Record Dates: First submitted 2015-07-24; First posted 2015-07-28 (Estimated); Results first posted 2019-02-11 (Actual); Last update posted 2019-02-11 (Actual); Status verified 2019-02

CONDITIONS: Uterine Cervical Neoplasms
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — technetium-diethylenetriaminepentaacetic acid-mannosyl-dextran

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tc99m tilmanocept (Experimental): 2 mCi (74 MBq), 50 ug of Tc99M tilmanocept single administration
  Interventions: Drug: Tc99m tilmanocept

INTERVENTIONS:
Drug: Tc99m tilmanocept — A single dose of 2 mCi (74 MBq) and 50 ug of Tc99m tilmanocept administered peritumorally no more than 20 hours before surgery
  Other Names: Lymphoseek

SUMMARY:
Prospective, open-label, within-patient, multi-center study of Lymphoseek in the detection of lymph nodes in subjects with known cancer of the cervix. All subjects will receive a single dose of 50 µg Lymphoseek radiolabeled with 2 mCi (74 MBq) Tc 99m.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided written informed consent with HIPAA authorization
* Has cervical cancer and is a candidate for surgical intervention, with lymph node dissection being a part of the surgical plan.
* Is at least 18 years of age at the time of consent
* Has an ECOG performance status of Grade 0 to 2
* Has the following International Federation of Gynecology and Obstetrics (FIGO) IA2-IIA1staging. Subjects with a single enlarged/suspicious node on PET/CT will still be considered eligible as consistent with FIGO guidelines.
* If of childbearing potential, the subject has a negative pregnancy test within 48 hours before administration of Lymphoseek, has been surgically sterilized, or has been postmenopausal for at least 1 year

Exclusion Criteria:

* The subject has had preoperative chemotherapy, immunotherapy, or radiation therapy within the 30 days prior to Lymphoseek administration
* Has had previous surgery or radiation to node basins that would be involved in the ILM procedure
* Has a known allergy to dextran
* Is breast-feeding or pregnant
* Before the administration of Lymphoseek, has received any radiopharmaceutical within 7 radioactive half-lives of that radiopharmaceutical
* Is scheduled for surgery and/or another invasive procedure other than the primary surgical intervention within the 3 days after Lymphoseek administration
* Has received an investigational product within the 30 days prior to Lymphoseek administration

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-01; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Blue, MD, Study Director — Cardinal Health 414, LLC
Locations (4):
- United States (4):
  - University of California, San Diego, La Jolla, California
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - The University of Texas M.D. Anderson Cancer Center, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tc99m Tilmanocept
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Tc99m Tilmanocept: Enrolled subjects who were administered any injection of Tc99m tilmanocept.
Arm/Group | Tc99m Tilmanocept
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.53 (7.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 18
ECOG Status [Count of Participants; unit: Participants] — Grade 0: Fully active (better outcome) Grade 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature Grade 2: Ambulatory and capable of all self-care but unable to carry out any work activities Grade 3: Capable of only limited self-care Grade 4: Completely disabled. Cannot carry on any self-care. Grade 5: Dead (worse outcome)
  Participants
    0 | 18
    1 | 0
    2 | 0
    3 | 0
    4 | 0
    5 | 0

OUTCOME MEASURES:

1. Primary Outcome: Per-subject False Negative Rate
Description: Proportion of subjects with pathologically negative Lymphoseek-identified SLNs and at least one pathologically positive non-SLN
Time Frame: 1 day
Population: Participants receiving a single dose of 50 µg Lymphoseek radiolabeled with 2 mCi (74 MBq) Tc 99m for whom at least one lymph node was removed with histopathology available
Measure: Number (95% Confidence Interval); unit: Proportion of Participants
Groups:
- Intent-To-Treat: 2 mCi (74 MBq), 50 ug of Tc99M tilmanocept single administration
  Tc99m tilmanocept: A single dose of 2 mCi (74 MBq) and 50 ug of Tc99m tilmanocept administered peritumorally no more than 20 hours before surgery
Arm/Group | Intent-To-Treat
Number analyzed (Participants) | 18
Proportion of Participants | .333 [.0084 to .9057]

2. Secondary Outcome: Per-subject Sensitivity
Description: Proportion of subjects with at least one pathologically positive Lymphoseek-identified SLN that have at least one pathologically positive lymph node
Time Frame: 1 day
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Intent-To-Treat
Number analyzed (Participants) | 18
Proportion of participants | .667 [.0942 to .9916]

3. Secondary Outcome: Per-subject Negative Predictive Value
Description: Proportion of subjects with pathologically negative Lymphoseek-identified SLN(s) with no pathologically positive lymph nodes
Time Frame: 1 day
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Intent-To-Treat
Number analyzed (Participants) | 18
Proportion of participants | .9375 [.6977 to .9984]

4. Secondary Outcome: Per-subject Accuracy
Description: Proportion of subjects accurately indentified by Lymphoseek
Time Frame: 1 day
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Intent-To-Treat
Number analyzed (Participants) | 18
Proportion of participants | .9444 [.7271 to .9986]

5. Secondary Outcome: Proportion of Lymph Nodes Identified Intraoperatively by a Dye That Are Also Identified by Lymphoseek
Time Frame: 1 day
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Proportion of Condordant Nodes
Units Other Than Participants: Dye Positive Nodes
Arm/Group | Intent-To-Treat
Number analyzed (Participants) | 18
Number analyzed (Dye Positive Nodes) | 41
Proportion of Condordant Nodes | .8049 [.6513 to .9118]

6. Secondary Outcome: Number of Lymph Nodes Per-subject Identified by Lymphoseek
Time Frame: 1 day
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Nodes Per Subject
Units Other Than Participants: Total Lymph Nodes
Arm/Group | Intent-To-Treat
Number analyzed (Participants) | 18
Number analyzed (Total Lymph Nodes) | 49
Nodes Per Subject | 2.72 [2.09 to 3.36]

7. Secondary Outcome: Number of Lymph Nodes Per-subject Identified by Other Dyes
Time Frame: 1 day
Measure: Mean (95% Confidence Interval); unit: Nodes Per Subject
Units Other Than Participants: Total Lymph Nodes
Arm/Group | Intent-To-Treat
Number analyzed (Participants) | 18
Number analyzed (Total Lymph Nodes) | 41
Nodes Per Subject | 2.41 [1.64 to 3.18]

8. Secondary Outcome: Per-subject Concordance
Description: Subjects whose lymph nodes were determined to be dye positive that were also identified by Lymphoseek
Time Frame: 1 day
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Proportion of Condordant Subjects
Units Other Than Participants: Dye Positive Nodes
Arm/Group | Intent-To-Treat
Number analyzed (Participants) | 18
Number analyzed (Dye Positive Nodes) | 15
Proportion of Condordant Subjects | 1.0 [.7819 to 1.0]

9. Secondary Outcome: Per-subject Reverse Concordance
Description: Number of subjects whose lymph nodes that were identified by Lymphoseek were also all identified by dye
Time Frame: 1 day
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Proportion of Reverse Condordant Subj.
Units Other Than Participants: Hot Positive Nodes
Arm/Group | Intent-To-Treat
Number analyzed (Participants) | 18
Number analyzed (Hot Positive Nodes) | 18
Proportion of Reverse Condordant Subj. | .8333 [.5858 to .9642]

10. Secondary Outcome: Incidence of Adverse Events
Time Frame: 7 days
Population: Enrolled subjects who were administered any injection of Tc99m tilmanocept.
Measure: Number; unit: Events
Groups:
- Tc99m Tilmanocept: Enrolled patients who were administered any injection of Lymphoseek.
Arm/Group | Tc99m Tilmanocept
Number analyzed (Participants) | 18
Events | 5

ADVERSE EVENTS:
Time Frame: Day of injection through 24 hours post injection
Arm/Group | Tc99m Tilmanocept
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 5/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tc99m Tilmanocept (N=18)
Headache (Nervous system disorders) | 1 (1) — Not related to Lymphoseek.
Pain in right arm (Musculoskeletal and connective tissue disorders) | 1 (1) — Not related to Lymphoseek.
Nausea (Gastrointestinal disorders) | 1 (1) — Not related to Lymphoseek.
Vaginal bleeding (Reproductive system and breast disorders) | 1 (1) — Not related to Lymphoseek.
Small amount of bleeding at 3:00 injection site (Injury, poisoning and procedural complications) | 1 (1) — Not related to Lymphoseek.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI shall not submit a publication to journals or professional societies without the prior written approval of the Sponsor.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-11-03): https://cdn.clinicaltrials.gov/large-docs/85/NCT02509585/Prot_SAP_000.pdf